CLINICAL TRIAL: NCT06986291
Title: Quantitative Assessment of Radiation-induced Toxicity of the Heart
Brief Title: Radiation-induced Toxicity of the Heart
Acronym: CorTox
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Principal Investigator, Prof. Esther Troost, Prof. Dr. med. Dr., Technische Universität Dresden
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STR-CorTox-2024
Record Dates: First submitted 2025-05-15; First posted 2025-05-23 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Non-small Cell Lung Cancer; Esophageal Cancer; Breast Cancer Female
Keywords: Non-small cell lung cancer; Esophageal cancer; Breast cancer; Cardiotoxicity; Radio(chemo)therapy; MRI; Cardiac function test; Omics analyses
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Esophageal Neoplasms; Breast Neoplasms; Cardiotoxicity | interventions — Diagnostic Imaging

STUDY DESIGN:
Intervention Model Description: There are two cohorts (patients with non-small cell lung or esophageal cancer; patients with breast cancer) but receiving the same intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic (Other): Patients with non-small cell lung or esophageal cancer (cohort 1) or with breat cancer (cohort 2)
  Interventions: Diagnostic Test: Imaging and biomarkers

INTERVENTIONS:
Diagnostic Test: Imaging and biomarkers — MR imaging of the heart, ECG and TTE measurements, blood sample

SUMMARY:
Late side effects in radio(chemo)therapy [R(CH)T] pose a critical limitation to patients' overall survival and quality of life. Even though toxicities of the heart are highly relevant for patients with cancer in the thoracic region, risk stratification models for these toxicities are lacking. In this study, liquid, functional and imaging biomarkers are being investigated for their use in prediction of cardiac toxicity following R(CH)T for patients with thoracic malignancies.

DETAILED DESCRIPTION:
79 patients with non-small cell lung or esophageal cancer, and 246 patients with breast cancer to be treated with curative R(CH)T at the University Hospital Carl Gustav Carus Dresden, Germany will be included in this investigation. Dosimetric parameters from the applied radiation treatment plans, magnetic-resonance-imaging, electrocardiography, transthoracic echocardiography as well as blood-biomarkers will be collected to determine their predictive power against the primary endpoint of cumulative grade ≥ 2 cardio-toxicity (Common Terminology Criteria for Adverse Events [CTCAE] v 5.0) 3-5 years after R(CH)T.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years old or older
* Patient's consent and written consent is available
* Patients with the non-small cell lung cancer or esophageal cancer or breast cancer who have an indication for intended curative radio(chemo)therapy (in the case of breast cancer inclusion of female patients only)

Exclusion Criteria:

* Patients who are not capable of giving consent
* Pregnant women
* Patients with contraindications for MRI examinations (pacemakers, defibrillators, neurostimulators, aneurysm clips, cochlear implants, permanent make-up, metal splinters or osseosynthetic implants)
* Patients with insufficient kidney function (glomerular filtration rate (GFR) of less than 30 ml/min)
* Patients with the aforementioned tumour entities for whom a palliative indication exists

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only female patients with breast cancer (cohort 2)
Enrollment: 325 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2034-12 (Estimated); Study Completion 2039-12 (Estimated)

PRIMARY OUTCOMES:
Cumulative cardio-toxicity after 1 or 5 years | 12 or 60 months after end of treatment
  Cumulative grade ≥ 2 cardio-toxicity (Common Terminology Criteria for Adverse Events [CTCAE] v 5.0) 1 years after R(CH)T in patients with non-small cell lung or esophageal cancer or 5 years after R(CH)T in patients with breast cancer

SECONDARY OUTCOMES:
Cumulative cardio-toxicity (early and late) | 3 months as well as 2, 3, 4, 5 and 10 years after end of treatment
  Cumulative grade ≥ 2 cardio-toxicity (Common Terminology Criteria for Adverse Events [CTCAE] v 5.0) 3 months as well as 2, 3, 4 or 5 years after R(CH)T and in addition 10 years after R(CH)T in patients with breast cancer only.

CONTACTS AND LOCATIONS:
Overall Officials: Esther G. C. Troost, Prof. Dr. med. Dr., Principal Investigator — Department of Radiotherapy and Radiation Oncology, Faculty of Medicine and University Hospital Carl Gustav Carus, TUD Dresden University of Technology, Dresden, Germany
Locations (1):
- University of Technology, University Hospital Carl Gustav Carus, Department of Radiation Therapy and Radiation Oncology, Dresden, Germany, Germany

IPD SHARING:
Plan to Share IPD: No